CLINICAL TRIAL: NCT05486000
Title: Evaluating the Safety and Efficacy of Atrial Shunt Implantation Systems for the Treatment of Patients With Chronic Left Heart Failure Prospective, Multicenter, Single-group Target Value Clinical Trials
Brief Title: To Assess the Safety and Efficacy of the Atrial Shunt Implant System in the Treatment of Patients With Chronic Left Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morningside (Nantong) Medical Co.,Ltd (Other)
Collaborators: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-ATRIAL SEPTAL-2022-01
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Left Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): This group contains patients with chronic left heart failure who are undergoing intervention in the atrial shunt implant system
  Interventions: Device: Atrial shunt implant system

INTERVENTIONS:
Device: Atrial shunt implant system — Patients with chronic left heart failure who meet the conditions of the clinical trial undergo interventional surgery with the "Atrial Shunt Implant System"

SUMMARY:
This trial is a prospective, multicenter, single-group target-value clinical trial in which patients with chronic left heart failure are planned to be recruited.

Using the atrial shunt implantation system developed and produced by Morningside (Nantong) Medical Device Co., Ltd., the atrial septum is used to implant the instruments in the atrial septum.

to verify the safety and efficacy of the atrial shunt implant system for the treatment of patients with chronic left heart failure.

DETAILED DESCRIPTION:
This trial will be carried out in a number of clinical trial institutions in China, and a total of 120 subjects are planned to be included, and all subjects are in progress The single group was registered and surgically treated with an atrial shunt implant system and within 7 days of surgery or at the time of discharge, 30 days after surgery Clinical follow-up was carried out at 3 months after surgery, 6 months after surgery, and 12 months after surgery, followed by data collection, evaluation and statistics Analysis and 12 months of phased clinical summary submitted registration application, on this basis, complete 2 years, 3 years of long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Consistently stable GDMT (Guidelines for Guiding Drugs) according to The Chinese Guidelines for the Diagnosis and Treatment of Heart Failure 2018 Treatment) heart failure for patients with chronic left heart failure who are still symptomatic for at least 1 month;
3. History of hospital admission to heart failure in the past 12 months, serum BNP or NT-proBNP liters" within 6 months High (BNP in sinus rhythm patients> 70 pg/ml, atrial fibrillation patients > 200 pg/ml, or sinus rhythm patients NT-proBNP"> 200 pg/ml, patients with atrial fibrillation >600 pg/ml);
4. Cardiac catheterization measures resting mean lung capillary wedge pressure PCWP or left atrial pressure LAP≥15 mmHg,And the difference between the RAP order of pulmonary capillary wedge pressure PCWP and right atrial pressure is ≥ 5 mmHg；
5. Cardiac Function Classification (NYHA) Grade II-IV;
6. The patient or his/her guardian can understand the purpose of the study, voluntarily participate and sign a written informed consent form, which is acceptable Patients followed up； -

Exclusion Criteria:

1. Primary organic valvular disease and severe coronary artery disease requiring revascularization that are currently indicated for surgical intervention Changes, heart-related diseases indicated for pacemaker implantation treatment;
2. Pulmonary hypertension (pulmonary vascular resistance PVR>4WoodsUnits);
3. History of myocardial infarction or heart treatment surgery within three months;
4. Patients with infective endocarditis or ultrasound findings of thrombosis or vegetations in the heart;
5. Anatomical abnormalities that make surgery unfinished or anatomically unsuitable for surgery;
6. Life expectancy < 12 months;
7. History of stroke, transient cerebral ischemia, deep vein thrombosis or pulmonary embolism in the past 6 months;
8. Pregnant or lactating women, or persons with family planning in the next year;
9. Subjects whose judgement of poor compliance and who were unable to complete the study as required; -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The clinical treatment success rate was 12 months after operation | Twelve months after surgery
  Death and heart failure-related rehospitalization were avoided 12 months after surgery

SECONDARY OUTCOMES:
Instrument success rate | Intraoperative
  The diverter was successfully implanted, the morphology was normal, and the conveyor system was successfully withdrawn
Surgical success rate | Immediately after surgery
  On the basis of the success of the instrument, ultrasound is seen in simple left-to-right shunting immediately after surgery
6 minutes walking distance change | Preoperative screening ，30 days, 3 months, 6 months, 1 year after surgery 30 days, 3 months, 6 months, 1 year, 2 years, 3 years after surgery
  The participants were assessed at the appropriate follow-up site
New York Cardiac Function Grading NYHA | Preoperative screening ，30 days, 3 months, 6 months, 1 year, 2 years, 3 years after surgery
  New York Cardiac Function Grading NYHA is divided into four levels, which are determined according to the clinical presentation of the patient, and the higher the level, the more severe the symptoms of heart failure
Kansas City Cardiomyopathy Quality of Life Scale KCCQ Changes | Preoperative screening ，30 days, 3 months, 6 months, 1 year after surgery
  Kansas City Cardiomyopathy Quality of Life Scale KCCQ Changes consisted of a total of 23 items with a score between 0-100, with higher scores indicating less adverse effects of heart failure on a patient's quality of life
NT-proBNP or BNP variation | Preoperative screening ，Before discharge, 30 days after surgery, 3 months, 6 months, 1 year
  Corresponding follow-up sites are obtained by laboratory blood tests
Probability of postoperative echocardiographic changes | During surgery, before discharge, 30 days after surgery, 3 months, 6 months, 1 year
  Obtained through instrumentation inspection
Incidence of device-related serious adverse events | 30 days after surgery
  Serious adverse events related to the instrument that occur after the implantation of the instrument, such as the shedding of the instrument, embolism, causing damage to the mitral or tricuspid valve, causing severe arrhythmias, infectious endocarditis, any need to re-operate the instrument to remove the instrument, etc
Serious adverse events and incidence of adverse events | Intraoperative complications, 30 days before discharge, 3 months, 6 months, 1 year, 2 years, 3 years
  Events that occur during clinical trials that result in death or serious deterioration of health status, as well as the probability of adverse medical events that occur after a subject is treated with a trial product

CONTACTS AND LOCATIONS:
Overall Officials: yan wang, dean, Principal Investigator — Xiamen Cardiovascular Hospital, Xiamen University
Locations (1):
- Atrial shunt implant system, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Result] Hao G, Wang X, Chen Z, Zhang L, Zhang Y, Wei B, Zheng C, Kang Y, Jiang L, Zhu Z, Zhang J, Wang Z, Gao R; China Hypertension Survey Investigators. Prevalence of heart failure and left ventricular dysfunction in China: the China Hypertension Survey, 2012-2015. Eur J Heart Fail. 2019 Nov;21(11):1329-1337. doi: 10.1002/ejhf.1629. PMID 31746111
- [Result] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Am Coll Cardiol. 2017 Aug 8;70(6):776-803. doi: 10.1016/j.jacc.2017.04.025. Epub 2017 Apr 28. No abstract available. PMID 28461007
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Zhang Y, Zhang J, Butler J, Yang X, Xie P, Guo D, Wei T, Yu J, Wu Z, Gao Y, Han X, Zhang X, Wen S, Anker SD, Filippatos G, Fonarow GC, Gan T, Zhang R; China-HF Investigators. Contemporary Epidemiology, Management, and Outcomes of Patients Hospitalized for Heart Failure in China: Results From the China Heart Failure (China-HF) Registry. J Card Fail. 2017 Dec;23(12):868-875. doi: 10.1016/j.cardfail.2017.09.014. Epub 2017 Oct 10. PMID 29029965
- [Result] Shah SJ, Borlaug BA, Kitzman DW, McCulloch AD, Blaxall BC, Agarwal R, Chirinos JA, Collins S, Deo RC, Gladwin MT, Granzier H, Hummel SL, Kass DA, Redfield MM, Sam F, Wang TJ, Desvigne-Nickens P, Adhikari BB. Research Priorities for Heart Failure With Preserved Ejection Fraction: National Heart, Lung, and Blood Institute Working Group Summary. Circulation. 2020 Mar 24;141(12):1001-1026. doi: 10.1161/CIRCULATIONAHA.119.041886. Epub 2020 Mar 23. PMID 32202936
- [Result] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822
- [Result] Sondergaard L, Reddy V, Kaye D, Malek F, Walton A, Mates M, Franzen O, Neuzil P, Ihlemann N, Gustafsson F. Transcatheter treatment of heart failure with preserved or mildly reduced ejection fraction using a novel interatrial implant to lower left atrial pressure. Eur J Heart Fail. 2014 Jul;16(7):796-801. doi: 10.1002/ejhf.111. Epub 2014 Jun 24. PMID 24961390
- [Result] Malek F, Neuzil P, Gustafsson F, Kaye DM, Walton A, Mates M, Sondergaard L, Ihlemann N, Mariani JA, Reddy V. Clinical outcome of transcatheter treatment of heart failure with preserved or mildly reduced ejection fraction using a novel implant. Int J Cardiol. 2015;187:227-8. doi: 10.1016/j.ijcard.2015.03.198. Epub 2015 Mar 18. No abstract available. PMID 25841123
- [Result] Hasenfuss G, Hayward C, Burkhoff D, Silvestry FE, McKenzie S, Gustafsson F, Malek F, Van der Heyden J, Lang I, Petrie MC, Cleland JG, Leon M, Kaye DM; REDUCE LAP-HF study investigators. A transcatheter intracardiac shunt device for heart failure with preserved ejection fraction (REDUCE LAP-HF): a multicentre, open-label, single-arm, phase 1 trial. Lancet. 2016 Mar 26;387(10025):1298-304. doi: 10.1016/S0140-6736(16)00704-2. PMID 27025436
- [Result] Kaye DM, Hasenfuss G, Neuzil P, Post MC, Doughty R, Trochu JN, Kolodziej A, Westenfeld R, Penicka M, Rosenberg M, Walton A, Muller D, Walters D, Hausleiter J, Raake P, Petrie MC, Bergmann M, Jondeau G, Feldman T, Veldhuisen DJ, Ponikowski P, Silvestry FE, Burkhoff D, Hayward C. One-Year Outcomes After Transcatheter Insertion of an Interatrial Shunt Device for the Management of Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2016 Dec;9(12):e003662. doi: 10.1161/CIRCHEARTFAILURE.116.003662. PMID 27852653
- [Result] Shah SJ, Feldman T, Ricciardi MJ, Kahwash R, Lilly S, Litwin S, Nielsen CD, van der Harst P, Hoendermis E, Penicka M, Bartunek J, Fail PS, Kaye DM, Walton A, Petrie MC, Walker N, Basuray A, Yakubov S, Hummel SL, Chetcuti S, Forde-McLean R, Herrmann HC, Burkhoff D, Massaro JM, Cleland JGF, Mauri L. One-Year Safety and Clinical Outcomes of a Transcatheter Interatrial Shunt Device for the Treatment of Heart Failure With Preserved Ejection Fraction in the Reduce Elevated Left Atrial Pressure in Patients With Heart Failure (REDUCE LAP-HF I) Trial: A Randomized Clinical Trial. JAMA Cardiol. 2018 Oct 1;3(10):968-977. doi: 10.1001/jamacardio.2018.2936. PMID 30167646
- [Result] Amat-Santos IJ, Bergeron S, Bernier M, Allende R, Barbosa Ribeiro H, Urena M, Pibarot P, Verheye S, Keren G, Yaacoby M, Nitzan Y, Abraham WT, Rodes-Cabau J. Left atrial decompression through unidirectional left-to-right interatrial shunt for the treatment of left heart failure: first-in-man experience with the V-Wave device. EuroIntervention. 2015 Jan;10(9):1127-31. doi: 10.4244/EIJY14M05_07. PMID 24832489
- [Result] Del Trigo M, Bergeron S, Bernier M, Amat-Santos IJ, Puri R, Campelo-Parada F, Altisent OA, Regueiro A, Eigler N, Rozenfeld E, Pibarot P, Abraham WT, Rodes-Cabau J. Unidirectional left-to-right interatrial shunting for treatment of patients with heart failure with reduced ejection fraction: a safety and proof-of-principle cohort study. Lancet. 2016 Mar 26;387(10025):1290-7. doi: 10.1016/S0140-6736(16)00585-7. PMID 27025435
- [Result] Rodes-Cabau J, Bernier M, Amat-Santos IJ, Ben Gal T, Nombela-Franco L, Garcia Del Blanco B, Kerner A, Bergeron S, Del Trigo M, Pibarot P, Shkurovich S, Eigler N, Abraham WT. Interatrial Shunting for Heart Failure: Early and Late Results From the First-in-Human Experience With the V-Wave System. JACC Cardiovasc Interv. 2018 Nov 26;11(22):2300-2310. doi: 10.1016/j.jcin.2018.07.001. Epub 2018 Nov 1. PMID 30391390
- [Result] Guimaraes L, Bergeron S, Bernier M, Rodriguez-Gabella T, Del Val D, Pibarot P, Eigler N, Abraham WT, Rodes-Cabau J. Interatrial shunt with the second-generation V-Wave system for patients with advanced chronic heart failure. EuroIntervention. 2020 Mar 20;15(16):1426-1428. doi: 10.4244/EIJ-D-19-00291. No abstract available. PMID 31422927
- [Result] Patel MB, Samuel BP, Girgis RE, Parlmer MA, Vettukattil JJ. Implantable atrial flow regulator for severe, irreversible pulmonary arterial hypertension. EuroIntervention. 2015 Oct;11(6):706-9. doi: 10.4244/EIJY15M07_08. PMID 26477643
- [Result] Rajeshkumar R, Pavithran S, Sivakumar K, Vettukattil JJ. Atrial septostomy with a predefined diameter using a novel occlutech atrial flow regulator improves symptoms and cardiac index in patients with severe pulmonary arterial hypertension. Catheter Cardiovasc Interv. 2017 Dec 1;90(7):1145-1153. doi: 10.1002/ccd.27233. Epub 2017 Sep 1. PMID 28862384
- [Result] Paitazoglou C, Ozdemir R, Pfister R, Bergmann MW, Bartunek J, Kilic T, Lauten A, Schmeisser A, Zoghi M, Anker S, Sievert H, Mahfoud F. The AFR-PRELIEVE trial: a prospective, non-randomised, pilot study to assess the Atrial Flow Regulator (AFR) in heart failure patients with either preserved or reduced ejection fraction. EuroIntervention. 2019 Aug 29;15(5):403-410. doi: 10.4244/EIJ-D-19-00342. PMID 31130524
- [Result] Paitazoglou C, Bergmann MW, Ozdemir R, Pfister R, Bartunek J, Kilic T, Lauten A, Schmeisser A, Zoghi M, Anker SD, Sievert H, Mahfoud F; AFR-PRELIEVE Investigators. One-year results of the first-in-man study investigating the Atrial Flow Regulator for left atrial shunting in symptomatic heart failure patients: the PRELIEVE study. Eur J Heart Fail. 2021 May;23(5):800-810. doi: 10.1002/ejhf.2119. Epub 2021 Mar 5. PMID 33555114
- See also: Guidelines for the diagnosis and treatment of heart failure — http://www.escardio.org/Guidelines/Clinical-Practice-Guidelines/Acute-and-Chronic-Heart-Failure